CLINICAL TRIAL: NCT00627861
Title: Renin System Responses to Combined Renin Inhibition and Beta Adrenergic Blockade
Brief Title: Combined Renin Inhibition/Beta-blockade
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The renin laboratory used in the study is no longer available.
Sponsor: The Rogosin Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0712009564
Record Dates: First submitted 2008-02-24; First posted 2008-03-04 (Estimated); Results first posted 2011-09-28 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aliskiren and metoprolol succinate (Experimental)
  Interventions: Drug: Aliskiren; Drug: Extended-release metoprolol

INTERVENTIONS:
Drug: Aliskiren — 150mg orally daily for 6 weeks. Dose may increase to 300mg orally daily dependent upon blood pressure parameters set by the protocol.
  Other Names: Tekturna
Drug: Extended-release metoprolol — 50mg orally daily for 1 week, dose will increase to 100mg orally daily or decrease to 25mg daily for a second week dependent upon blood pressure parameters set by the protocol. Subjects will take metoprolol for a total of 2 weeks, then be tapered off of it over 5-7 days.
  Other Names: Toprol-XL

SUMMARY:
Antihypertensive drug treatment is effective in only about 50% of patients. One mechanism responsible for treatment failure is a drug related stimulation of the renin-angiotension-aldosterone-system (RAAS). Several classes of medications that treat hypertension by blocking the RAAS system have been developed. However, the kidney responds to these drug treatments by producing greater amounts of renin. This high level of renin can reduce the effectiveness of some of these medications, ultimately causing the blood pressure to rise. This is one reason why blood pressure can be difficult to control in a certain percentage of patients.

The hypothesis to be tested in the proposed study is that beta-adrenergic blockade (β-blockade), when superimposed upon aliskiren, a drug that competitively inhibits plasma renin activity (PRA) but stimulates the release of renin by the kidneys (plasma renin concentration [PRC]), can suppress the reactive increase in PRC that occurs during aliskiren monotherapy.

The primary aim of this study is to measure plasma renin concentration (PRC) and plasma renin activity (PRA) levels during renin inhibition with aliskiren and combined renin inhibition/β-blocker treatment to determine whether the addition of a β-blocker attenuates the rise in plasma renin concentration (PRC). A secondary aim is to determine whether combined treatment further suppresses PRA and blood pressure.

DETAILED DESCRIPTION:
The renin-angiotensin-aldosterone system (RAAS) plays a central role in the maintenance of normal blood pressure (BP) homeostasis. Derangements in the regulation of this system, predominantly due to the failure to appropriately suppress renin secretion by the kidney, contribute to the pathogenesis of hypertension and its cardiovascular, renal and cerebrovascular complications.

Several classes of antihypertensive medications that interrupt the RAAS have been developed. These include agents that block angiotensin II (Ang II) binding to the AT1 receptor (Ang II receptor blockers [ARB]), inhibit conversion of Ang I to Ang II (angiotensin converting enzyme [ACE] inhibitors), and suppress renal secretion of renin (beta-adrenergic receptor blocker). These agents effectively lower BP, particularly in the hypertensive patient with an unsuppressed plasma renin activity (PRA) level, and significantly improve survival in cardiovascular diseases in which PRA levels are often elevated (e.g., heart failure, myocardial infarction).

Renin secretion is regulated, in part, by feedback inhibition due to Ang II binding to the juxtaglomerular cell (JG). Interruption of Ang II generation or its receptor binding during treatment with an ACE inhibitor or ARB, respectively, stimulates renin secretion because feedback inhibition is attenuated and renal perfusion pressure is reduced. The consequent, reactive rise in PRA that occurs during treatment with these drugs can limit their antihypertensive efficacy because Ang I and subsequently, Ang II levels increase.

These observations reinforce the theoretical and practical importance of pharmacologic suppression of renin secretion to prevent the reactive rise in PRA that occurs during treatment with ACE inhibitors and ARBs. β-blockers suppress renin secretion by inhibiting β1-adrenergic receptors located on JG cells. PRA and Ang II levels are highly correlated and these decrease commensurately during treatment with a β-blocker.

Aliskiren is an orally active, non-peptide renin inhibitor. Its antihypertensive efficacy is due to the competitive antagonism of the renin-mediated conversion of angiotensinogen to Ang I. During aliskiren treatment, PRA and Ang II levels decrease significantly. Unlike β-blockade, in which the PRA level decreases as a consequence of reduced renal secretion of renin, aliskiren treatment decreases PRA in response to the direct, competitive inhibition of renin. Although PRA decreases, the aliskiren-mediated decrease in plasma Ang II level stimulates renal renin secretion. Therefore, although aliskiren and β-blockers both decrease PRA levels, they have divergent effects on the plasma concentration of renin (PRC): β-blockers decrease it and aliskiren increases it. The reactive rise in PRC has potential implications regarding the antihypertensive efficacy of aliskiren - high PRC levels theoretically can overcome the competitive inhibition of renin by aliskiren, thereby increasing PRA, Ang II, and BP.

Aliskiren has been studied as monotherapy and in combination with other antihypertensive drugs, including hydrochlorothiazide, valsartan, and amlodipine. It has not been studied in the presence of a β-blocker. Proposals for future studies include pursuing whether or not there are hypertensives who are resistant to aliskiren, what the mechanism(s) is for the resistance and ways to overcome the resistance.

This is a prospective, open-label study of the effect of the sequential addition of a β-blocker (extended release metoprolol) to aliskiren on the levels of plasma renin activity and plasma renin concentration in subjects with uncomplicated hypertension.

ELIGIBILITY:
Inclusion Criteria:

Twenty subjects with a history of hypertension with the following inclusion criteria will be enrolled:

* Age 18-80 years
* Stage 1 (systolic 140-159 mm Hg or diastolic 90-99 mmHg) or Stage 2 (systolic >160 mm Hg or diastolic >100 mmHg) or current treatment with antihypertensive medication.
* PRA ≥0.65 ng/ml/h. If PRA is below this level during the screening period, due to treatment with a beta-blocker or central α2-receptor agonist, the subject may be enrolled and the PRA level re-checked after treatment is tapered off.

Exclusion Criteria:

* History of diabetes requiring pharmacologic treatment with an oral or parenteral hypoglycemic agent, including insulin
* TIA, stroke or myocardial infarction
* History of asthma or COPD
* Cockcroft Gault estimated GFR <60 ml/min/1.73 m2
* Previous adverse events during treatment with a β-blocker or aliskiren
* ALT level twice normal
* Secondary forms of hypertension (e.g., renovascular, primary aldosteronism)
* PRA<0.65 ng/ml/h after discontinuation of antihypertensive medication
* Systolic BP>180 mm Hg, diastolic BP>105 mm Hg
* Pregnant or breastfeeding, or planning pregnancy during the study period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon D Blumenfeld, M.D., Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

REFERENCES:
- [Background] Staessen JA, Li Y, Richart T. Oral renin inhibitors. Lancet. 2006 Oct 21;368(9545):1449-56. doi: 10.1016/S0140-6736(06)69442-7. PMID 17055947
- [Result] Nussberger J, Wuerzner G, Jensen C, Brunner HR. Angiotensin II suppression in humans by the orally active renin inhibitor Aliskiren (SPP100): comparison with enalapril. Hypertension. 2002 Jan;39(1):E1-8. doi: 10.1161/hy0102.102293. PMID 11799102
- [Result] Sealey JE, Laragh JH. Aliskiren, the first renin inhibitor for treating hypertension: reactive renin secretion may limit its effectiveness. Am J Hypertens. 2007 May;20(5):587-97. doi: 10.1016/j.amjhyper.2007.04.001. PMID 17485026
- [Result] Oparil S, Yarows SA, Patel S, Fang H, Zhang J, Satlin A. Efficacy and safety of combined use of aliskiren and valsartan in patients with hypertension: a randomised, double-blind trial. Lancet. 2007 Jul 21;370(9583):221-229. doi: 10.1016/S0140-6736(07)61124-6. PMID 17658393
- [Result] Blumenfeld JD, Sealey JE, Mann SJ, Bragat A, Marion R, Pecker MS, Sotelo J, August P, Pickering TG, Laragh JH. Beta-adrenergic receptor blockade as a therapeutic approach for suppressing the renin-angiotensin-aldosterone system in normotensive and hypertensive subjects. Am J Hypertens. 1999 May;12(5):451-9. doi: 10.1016/s0895-7061(99)00005-9. PMID 10342782

RESULTS

PARTICIPANT FLOW:
Groups:
- Aliskiren and Metoprolol: Aliskiren was administered for 4 weeks and then Metoprol was added for 2 additional weeks of treatment.
Period: Overall Study
Arm/Group | Aliskiren and Metoprolol
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Aliskiren and Metoprolol
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Plasma Renin Concentration
Time Frame: 5th, 6th, 7th, 9th, 10th, 11th, 12th weeks
Measure: Number; unit: pg/mL
Arm/Group | Aliskiren and Metoprolol
Number analyzed (Participants) | 1
pg/mL
  Week 5 | 16.5
  Week 6 | 13.5
  Week 7 | 20.5
  Week 9 | 22
  Week 10 | 2.7
  Week 11 | 4.4
  Week 12 | 3.2

2. Secondary Outcome: Plasma Renin Activity
Description: The blood test, plasma renin activity or PRA, is being measured during the visits outlined.
Time Frame: screening, 4th, 6th, 7th, 9th, 10th, 11th, 12th weeks
Measure: Number; unit: ng/mL/h
Groups:
- Aliskiren and Metoprolol: Aliskiren was administered for 4 weeks and then Metoprol was added for an additional 2 weeks.
Arm/Group | Aliskiren and Metoprolol
Number analyzed (Participants) | 1
ng/mL/h
  Screening | 2.07
  Week 4 | 1.22
  Week 6 | 0.28
  Week 7 | 0.18
  Week 9 | 0.28
  Week 10 | 0.07
  Week 11 | 0.03
  Week 12 | 0.06

3. Secondary Outcome: Blood Pressure
Time Frame: all visits (weekly for 12 weeks)
Measure: Number; unit: mm Hg
Arm/Group | Aliskiren and Metoprolol
Number analyzed (Participants) | 1
mm Hg
  Week 1-Systolic | 146
  Week 1-Diastolic | 64
  Week 2-Systolic | 144
  Week 2-Diastolic | 88
  Week 3-Systolic | 148
  Week 3-Diastolic | 90
  Week 4-Systolic | 148
  Week 4-Diastolic | 92
  Week 5-Systolic | 156
  Week 5-Diastolic | 92
  Week 6-Systolic | 150
  Week 6-Diastolic | 84
  Week 7-Systolic | 157
  Week 7-Diastolic | 89
  Week 8-Systolic | 147
  Week 8-Diastolic | 76
  Week 9-Systolic | 129
  Week 9 -Diastolic | 94
  Week 10-Systolic | 139
  Week 10-Diastolic | 79
  Week 11-Systolic | 170
  Week 11-Diastolic | 90
  Week 12-Systolic | 146
  Week 12-Diastolic | 78

ADVERSE EVENTS:
Arm/Group | Aliskiren and Metoprolol
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aliskiren and Metoprolol (N=1)
Leukocytosis (Immune system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes